CLINICAL TRIAL: NCT06411964
Title: Does Galactooligosaccharide Supplementation Improve Markers of Skeletal Muscle Health in Elderly Individuals?
Brief Title: Galactooligosaccharide and Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Adam Collins, Principal Investigator, University of Bath
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 239308
Record Dates: First submitted 2024-05-07; First posted 2024-05-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Muscle Loss
Keywords: sarcopenia; physical function; aging; gut microbiome; prebiotic
MeSH Terms: conditions — Muscular Atrophy; Sarcopenia | interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GOS (Experimental): Galactooligosaccharide (GOS) is a prebiotic supplement. Taken once daily for the duration for the intervention
  Interventions: Dietary Supplement: Prebiotic
- Placebo (Placebo Comparator): Maltodextrin placebo taken once daily for the duration of the intervention
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Prebiotic — Commercially available supplement (Bimuno)
  Arms: GOS
Dietary Supplement: Placebo control — maltodextrin control supplement
  Arms: Placebo

SUMMARY:
Sarcopenia is a progressive muscle disease, most commonly affecting older individuals, that is categorised by 1) low muscle strength, 2) low muscle quantity or quality, and 3) low physical performance. This disease has several negative implications for human health, including an increased risk of falls, fractures, mobility limitations, and mortality. Sarcopenia also imposes significant burden on healthcare systems. For example, it was estimated that a 10% reduction in the prevalence of sarcopenia would save the US healthcare system $1.1 billion per year. Strategies to reduce the incidence and severity of sarcopenia are therefore of great interest.

One potential cause for sarcopenia is long-term, low-level inflammation, which can occur for a number of reasons. One cause may relate to the intestinal wall becoming more susceptible to leaking of toxic particles. Evidence suggests that prebiotic supplementation can reduce this 'leakage'. Galactooligosaccharide (a prebiotic) has previously been shown to reduce inflammation in elderly individuals. The investigators hypothesise that galactooligosaccharide will improve physical function in the elderly indirectly via a reduction in inflammation.

This will be a randomised, placebo-controlled, double-blind, parallel study. 32 elderly individuals (65-85 years; mix of males and females) will be randomised to one of two groups, GOS or PLACEBO. The GOS group will supplement their diet with 2.9 g galactooligosaccharide per day for 16 weeks in the form of one sachet (3.65 g) of Bimuno® Daily.

The PLACEBO group will supplement with 3.65 g maltodextrin per day for 16 weeks. The study will involve one screening visit and two main trials (baseline and 16 weeks). For the main trials, participants will complete the short physical performance battery (SPPB) and handgrip strength test. In addition, participants will provide blood, urine and faecal samples, as well as a dual-energy x-ray absorptiometry (DEXA), and a peripheral quantitative computed tomography (pQCT) scan.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-85 years
* Able to rise from a chair without using arms

Exclusion Criteria:

* Use of products marketed as prebiotics, probiotics or synbiotics within 4 weeks prior to study entry (e.g., Yakult, Actimel, Activia, VSL#3, Kefir). Regular cheese or yogurt containing lactic acid bacteria are not an exclusion criterion

  * Systemic antibiotic or antimycotic treatment 6 weeks prior to study entry.
  * Following diets likely to affect study outcomes: e.g., low FODMAP, KETO/high-fat, gluten free/coeliac, paleo, weight loss, caloric restriction, low-carb, 5:2/whole day energy restriction, Atkins/high-protein, sugar-free, single-food, juicing/any day of juicing, any other restriction diet (e.g. very low calorie), or vegan diets (GOS is derived from cow's milk)
  * Meeting physical activity guidelines for older adults:
* Activities that improve strength, flexibility and balance at least two days per week
* At least 150 minutes of moderate-intensity activity, or 75 minutes of vigorous activity

  * Body mass loss of ≥ 5% in preceding 6 months
  * History of injury or surgery that would affect physical ability to undertake physical tests
  * History of gastrointestinal disease (e.g., inflammatory bowel disease, irritable bowel syndrome)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-10-06 (Estimated); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
Mid-thigh muscle cross sectional area | 16 weeks
  pQCT assessment of mid-thigh cross sectional area

SECONDARY OUTCOMES:
Short performance physical battery | 16 weeks
  composite test of balance, gait speed and chair stand tests where performance on each three tests scores of maximum of 4 points, combined to score a maximum of 12 points
Handgrip strength | 16 weeks
  dominant and non-dominant hand scores
appendicular lean mass/height^2 (kilograms/metres^2) | 16 weeks
  assessed via DEXA scan
gait speed | 16 weeks
  4m gait speed at usual walking pace (metres/second)
chair stand | 16 weeks
  5 time chair stand (seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Bath and NE Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No